CLINICAL TRIAL: NCT04133103
Title: A Prospective Study of Early Mobilisation in the Surgical Robot Assisted Spinal Surgery
Brief Title: Early Mobilisation in the Surgical Robot Assisted Spinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Wei Tian, director of spine department, Beijing Jishuitan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Jilunke201909-24
Record Dates: First submitted 2019-10-13; First posted 2019-10-21 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-10

CONDITIONS: Degenerative Disease; Fracture
Keywords: early mobilisation; robot; spine; enhanced recovery
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First ambulation at 24 hours after operation (No Intervention)
- First ambulation at 4 hours after operation (Experimental)
  Interventions: Procedure: first ambulation at 4 hour after operation

INTERVENTIONS:
Procedure: first ambulation at 4 hour after operation — Two groups were conducted for first ambulation at 4 or 24 hours aftër operation
  Arms: First ambulation at 4 hours after operation

SUMMARY:
In this study, patients who underwent lumbar spine surgery in our hospital were included. A prospective study was conducted to investigate the effects of early mobilisation on postoperative complications, functual outcomes and patient satisfaction after robotic assisted lumbar spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of degenerative diseases or spinal fracture
* single level instrumentation sugery
* sign informed consent

Exclusion Criteria:

* multilevel instrumentaion surgery
* diagnosis of severe osteoperosis (BMD < 60mg/cm3) by QCT
* coagulant function abnormality
* severe internal disease
* not suitable for inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-03-02 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | preoperative
  Low back pain and leg pain is an important sign and a frequent patient complaint. The VAS pain scoring standard (scores from 0 to 10) was as following: 0 means painless; 1-3 means mild pain that the patient could endure; 4-6 means patient was in pain that could be endured and be able to sleep; and 7-10 means patient had intense pain and was unable to tolerate the pain.
Visual Analogue Scale | 4 hours postoperatively
  Low back pain and leg pain is an important sign and a frequent patient complaint. The VAS pain scoring standard (scores from 0 to 10) was as following: 0 means painless; 1-3 means mild pain that the patient could endure; 4-6 means patient was in pain that could be endured and be able to sleep; and 7-10 means patient had intense pain and was unable to tolerate the pain.
Visual Analogue Scale | 24 hours postoperatively
  Low back pain and leg pain is an important sign and a frequent patient complaint. The VAS pain scoring standard (scores from 0 to 10) was as following: 0 means painless; 1-3 means mild pain that the patient could endure; 4-6 means patient was in pain that could be endured and be able to sleep; and 7-10 means patient had intense pain and was unable to tolerate the pain.
Visual Analogue Scale | 3 months postoepratively
  Low back pain and leg pain is an important sign and a frequent patient complaint. The VAS pain scoring standard (scores from 0 to 10) was as following: 0 means painless; 1-3 means mild pain that the patient could endure; 4-6 means patient was in pain that could be endured and be able to sleep; and 7-10 means patient had intense pain and was unable to tolerate the pain.

SECONDARY OUTCOMES:
Japanese Orthopedic Association | preoperative
  The Japanese Orthopedic Association score was used to evaluate the neurological function of patients with lumbar degeneration and treatment effectiveness. The highest possible total score from categories for a normal person is 29 points. Therefore, treatment improvement rate = [(post-treatment score - pre-treatment score) / (29 - pre-treatment score)] × 100%, and ≥75% means excellent; 50%-74% means good; 25%-49% means fair; 0-24% means poor.
Japanese Orthopedic Association | 3 months postoperatively
  The Japanese Orthopedic Association score was used to evaluate the neurological function of patients with lumbar degeneration and treatment effectiveness. The highest possible total score from categories for a normal person is 29 points. Therefore, treatment improvement rate = [(post-treatment score - pre-treatment score) / (29 - pre-treatment score)] × 100%, and ≥75% means excellent; 50%-74% means good; 25%-49% means fair; 0-24% means poor.
Oswestry Disability Index | preoperative
  The Oswestry Disability Index is one of the principal condition-speciﬁc outcome measures used in the management of spinal disorders. Rounding the percentage to a whole number is suggested for convenience. So the final score may be summarized as: [total score / (5 × number of questions answered)] × 100%. It is suggested rounding the percentage to a whole number for convenience. We defined that 0-20% means mild; 21%-40% means moderate; 41%-60% means severe; 61%-80% means very severe；80%-100% means patients very exaggerated symptoms.
Oswestry Disability Index | 3 months postoperatively
  The Oswestry Disability Index is one of the principal condition-speciﬁc outcome measures used in the management of spinal disorders. Rounding the percentage to a whole number is suggested for convenience. So the final score may be summarized as: [total score / (5 × number of questions answered)] × 100%. It is suggested rounding the percentage to a whole number for convenience. We defined that 0-20% means mild; 21%-40% means moderate; 41%-60% means severe; 61%-80% means very severe；80%-100% means patients very exaggerated symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Tian, Study Director — Beijng Jishuitan Hospital
Locations (1):
- Wei Tian, Beijing, China

IPD SHARING:
Plan to Share IPD: No